CLINICAL TRIAL: NCT02114905
Title: Dissemination of Comprehensive Behavioral Intervention for Tics (CBIT) to Occupational Therapists: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1208012814
Record Dates: First submitted 2014-02-06; First posted 2014-04-15 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Tourette Disorder; Chronic Tic Disorder
Keywords: Tourette's; Tic Disorder; CBIT; Dissemination; Occupational Therapist
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OTs Trained and Deliver CBIT (Experimental): CBIT certified clinicians will train OTs in delivering CBIT to affected youth. OTs will be supervised in the practice of CBIT with youth in the New York City and Birmingham areas. Pre- and post-treatment assessment measures will be collected from 16 families (8 from each site) to evaluate intervention acceptability, feasibility, and fidelity. Patient and parent satisfaction of CBIT-OT will also be documented.
  Interventions: Behavioral: OTs Trained and Deliver CBIT

INTERVENTIONS:
Behavioral: OTs Trained and Deliver CBIT — CBIT is a highly structured therapy that typically takes place on a weekly basis. The patient is taught to perform a specific behavior that makes the tic more difficult to do, as soon as the tic or urge appears. This "competing response" helps to reduce, and in some cases, even eliminate the tic. The functional intervention (FI), is based on the fact that certain situations or reactions to tics can make them worse than they might otherwise be. The goal of FI is to identify these situations and have the patient and family attempt to change them so the tics aren't made worse unnecessarily.
  Other Names: CBIT

SUMMARY:
Comprehensive Behavioral Intervention for Tics (CBIT) is an evidence based intervention for tic disorders. A recent scientific review of research priorities completed by the Tourette Syndrome Association recommended widespread dissemination of CBIT as an important next step in services delivery research. Given early evidence that occupational therapists can deliver CBIT effectively, a dissemination strategy using occupational therapists may improve accessibility to this treatment, at lower cost and with decreased stigma. Thus the goal of this study is to develop and test a training and dissemination model with occupational therapists (OTs) using an expert, multi-disciplinary team at Weill Cornell/New York Presbyterian Hospital (WC/NYPH) and University of Alabama at Birmingham (UAB). The investigators have adapted CBIT, the gold-standard behavioral intervention program for children with tic disorders (Woods et al, 2008a,b), for eventual use in OT programs across the country.

DETAILED DESCRIPTION:
CBIT training materials designed by the study team have been used to train occupational therapists (OTs) at WC/NYPH and UAB to deliver CBIT, and data has been collected to measure training acceptability.

OTs will be supervised in the practice of CBIT with youth in the New York City and Birmingham areas. Pre- and post-treatment assessment measures will be collected from 16 families (8 from each site) to evaluate intervention acceptability, feasibility, and fidelity. Patient and parent satisfaction of CBIT-OT will also be documented. The investigators will look within subjects to ascertain change in reported tic severity.

This study is designed to determine the feasibility and acceptability of treatment, feasibility of research design, as well as demonstrate the ability to disseminate the study protocol to a new care discipline in methodologically rigorous fashion across multiple sites.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-17
* Presence of motor and/or vocal tics for at least 6 months
* Tics are of at least moderate clinical severity as evidenced by a Clinical Global Impressions Severity (CGI-S) score of 4 or higher (tic symptoms clearly noticeable to family and occasionally to families and associated with at least some minimal level of distress and/or interference.
* IQ estimate of 70 or higher
* Comorbid disorder (e.g., ADHD, OCD,ODD) will be allowed provided that the tic symptoms are of primary concern to parents and comorbid symptoms are not of sufficient severity to require immediate treatment other than that provided by the current study.
* Pre-existing stable medication, tic or otherwise, will also be allowed provided the family agrees to refrain from med changes over the course of the study if at all possible.
* Sufficient command of the English language to comply with study protocol.

Exclusion Criteria:

* Free of PDD or other developmental disability

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2013-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Treatment Acceptability Questionnaire | One year
  OT's will fill out a questionnaire at the completion of the study regarding their assessment of the training module, training materials, and their comfortability and confidence delivering CBIT to children.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Bennett, PhD, Principal Investigator — Weill Medical College of Cornell University; Jan Rowe, OT, Study Chair — University of Alabama at Birmingham
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No